CLINICAL TRIAL: NCT05726318
Title: A Randomized Pilot and Feasibility Study of a cultuRE-Directed Approach to Urinary traCT Infection Symptoms in Older womeN: a Mixed Methods Evaluation - the REDUCTION Trial
Brief Title: Randomized Trial of Culture Directed Versus Empiric Antibiotics for Urinary Tract Infections in Older Women
Acronym: REDUCTION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Megan Bradley (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Megan Bradley, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY22060176; DK131273 (Other: NIDDK); R01DK131273 (NIH)
Record Dates: First submitted 2023-01-19; First posted 2023-02-13 (Actual); Results first posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: UTI
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Culture-directed antibiotic (Other): Participants will be directed to refrain from taking antibiotics until results of urine culture are reported, which is expected within 48-72h.
  Interventions: Drug: Antibiotics
- Empiric antibiotic (Active Comparator): Antibiotic Protocol. For participants in the empiric Rx arm, we will choose an antibiotic with consideration of patient reported allergies, current medications and current Infectious Disease Society of American (IDSA) guidelines. If there is a contraindication to the first antibiotic on the list they will progress to the next option until a suitable selection is achieved.
  Interventions: Drug: Antibiotics

INTERVENTIONS:
Drug: Antibiotics — Participants will be provided either nitrofurantoin 100 mg oral twice a day for 5 days, trimethoprim/sulfamethoxazole 875/125 oral twice a day for 3 days, fosfomycin 3g once oral, ciprofloxacin 250 mg oral twice a day for 5 days or cephalexin 500 mg oral twice a day for 5 days

SUMMARY:
To evaluate the feasibility of recruiting eligible subjects into a randomized trial of a culture-directed versus empiric antibiotic strategy for patient-reported urinary tract infection symptoms in older women and the adherence to study procedures.

DETAILED DESCRIPTION:
To evaluate A) the feasibility of recruiting eligible subjects into a randomized trial of a culture-directed versus empiric antibiotic strategy for patient-reported urinary tract infection (UTI) symptoms in older women and B) the adherence to study procedures. We will recruit and enroll women with a history of recurrent UTI (rUTI) from the Women's Center for Bladder and Pelvic Health and the University of Pittsburgh's Clinical and Translational Science Institute (CTSI) Pitt+Me® Research Registry. Once enrolled and randomized, women will be followed for a total of 28 days to document both clinical resolution at day 7 from symptom onset and adverse events. H1) Enrolling a total of 70 subjects in <1 year (at least 10% of eligible patients) will demonstrate feasibility of recruitment and H2) Documenting at least 70% patient compliance with study procedures will confirm patient adherence to study protocol. Exploratory Aim: To explore the safety of a culture-directed UTI treatment strategy and preliminary secondary outcomes of assigned treatments. H1) There will be an overall low number of adverse events and H2) Preliminary outcome data will help power future trial.

ELIGIBILITY:
Inclusion Criteria:

* Female biologic Sex
* Age ≥65 years old
* History of recurrent UTI per patient report of greater than 2 UTIs in the last 6 months or 3 UTIs in the last year
* Patient reported UTI defined as:

  * Dysuria, increased urinary urgency/frequency and/or suprapubic pain

Exclusion Criteria:

* Male biologic sex
* Age <65 years old
* History of augmentation cystoplasty or cystectomy
* Currently performing clean intermittent self-catheterization
* Current indwelling foley catheter
* Urinary tract instrumentation (i.e., cystourethroscopy, foley catheter placement) in the last 30 days
* Undergoing treatment for malignancy
* History of either confirmed or patient reported pyelonephritis and/or urosepsis
* Cirrhosis and/or end stage liver disease
* Chronic kidney disease with most recent estimated glomerular filtration rate <50 ml/min
* Dementia and/or currently reside in skilled nursing facility
* Current high-dose chronic steroids (>20mg/day of prednisone)
* Previous solid organ transplant
* Provider concern for pyelonephritis and/or sepsis (i.e., fevers)
* Unwilling or unable to comply with study procedures

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan S Bradley, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee Women's Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Will review each request individually and work with University of Pittsburgh Research Agreements to share.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year after completion
Access Criteria: unknown at this time

RESULTS

PARTICIPANT FLOW:
Groups:
- Empiric Antibiotic: Antibiotic Protocol. For participants in the empiric Rx arm, we will choose an antibiotic with consideration of patient reported allergies, current medications and current Infectious Disease Society of America (IDSA) guidelines. If there is a contraindication to the first antibiotic on the list they will progress to the next option until a suitable selection is achieved.
  Antibiotics: Participants will be provided either nitrofurantoin 100 mg oral twice a day for 5 days, trimethoprim/sulfamethoxazole 875/125 oral twice a day for 3 days, fosfomycin 3g once oral, ciprofloxacin 250 mg oral twice a day for 5 days or cephalexin 500 mg oral twice a day for 5 days
Period: Overall Study
Arm/Group | Culture-directed Antibiotic | Empiric Antibiotic
Started | 35 | 35
Completed | 31 | 31
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Empiric Antibiotic: Antibiotic Protocol. For participants in the empiric Rx arm, we will choose an antibiotic with consideration of patient reported allergies, current medications and current IDSA guidelines. If there is a contraindication to the first antibiotic on the list they will progress to the next option until a suitable selection is achieved.
  Antibiotics: Participants will be provided either nitrofurantoin 100 mg oral twice a day for 5 days, trimethoprim/sulfamethoxazole 875/125 oral twice a day for 3 days, fosfomycin 3g once oral, ciprofloxacin 250 mg oral twice a day for 5 days or cephalexin 500 mg oral twice a day for 5 days
- Total: Total of all reporting groups
Arm/Group | Culture-directed Antibiotic | Empiric Antibiotic | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.1 (7.1) | 75.7 (6.8) | 74.9 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 35 | 34 | 69
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 35 | 34 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Number of Participants with Diabetes Mellitus [Count of Participants; unit: Participants] | 5 | 6 | 11
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.5 (7.6) | 28.5 (6.1) | 29.5 (6.9)
Pelvic Floor Distress Inventory-20 [Mean (Standard Deviation); unit: units on a scale] — The Pelvic Floor Distress Inventory - Short Form 20 (PFDI-20) is a validated, patient-reported outcome measure that assesses symptom distress related to pelvic floor disorders. The PFDI-20 consists of 20 items divided into three subscales: Each item is scored from 0 to 4. Each subscale is scored by: Calculating the mean of the answered items in that subscale and multiplying the mean by 25. The total PFDI-20 score is the sum of the three subscale scores. Interpretation of Scores: Higher scores represent worse pelvic floor symptom distress.
  units on a scale | 137.9 (59.9) | 146.0 (68.0) | 142.0 (63.7)

OUTCOME MEASURES:

1. Primary Outcome: Eligible Subjects That Were Enrolled in the Study
Description: Number and proportion of eligible subjects that were enrolled in the study
Time Frame: Through study completion, an average of 17.5 months
Population: There were 103 eligible participants in the study time frame
Measure: Count of Participants; unit: Participants
Groups:
- Overall Number and Proportion of Eligible Subjects That Were Enrolled in the Study: Overall number and proportion of eligible subjects that were enrolled in the study
Arm/Group | Overall Number and Proportion of Eligible Subjects That Were Enrolled in the Study
Number analyzed (Participants) | 103
Participants | 70

2. Secondary Outcome: Number of Persons That Were Screened for Participation
Description: Overall number of persons that were screened for participation
Time Frame: Through study completion, an average of 17.5 months
Measure: Count of Participants; unit: Participants
Groups:
- Number of Subjects That Were Screened for Participation: Number of subjects that were screened for participation
Arm/Group | Number of Subjects That Were Screened for Participation
Number analyzed (Participants) | 131
Participants | 131

3. Secondary Outcome: Proportion of Persons Screened Who Met Inclusion/Exclusion Criteria
Description: Number of person screened who met include/exclusion criteria divided by number participants screened
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Groups:
- Number and Proportion of Subjects Screened Who Met Inclusion/Exclusion Criteria: Number and proportion of subjects screened who met inclusion/exclusion criteria
Arm/Group | Number and Proportion of Subjects Screened Who Met Inclusion/Exclusion Criteria
Number analyzed (Participants) | 131
Participants | 103

4. Secondary Outcome: Proportion of Persons Screened Who Declined Participation or Were Ineligible
Description: Number of person screened who declined or were ineligible divided by number participants screened
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Groups:
- Proportion of Persons Screened Who Declined Participation or Were Ineligible: Number of people screened who ultimately declined participation or were ineligible
Arm/Group | Proportion of Persons Screened Who Declined Participation or Were Ineligible
Number analyzed (Participants) | 131
Participants | 43

5. Secondary Outcome: Proportion of Participants Enrolled Who Completed the Study
Description: Number of persons enrolled who completed the study (at least one follow-up questionnaire and completed the day 28 questionnaire) divided by number participants enrolled
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Culture-directed Antibiotic | Empiric Antibiotic
Number analyzed (Participants) | 35 | 35
Participants | 30 | 31
Statistical Analysis 1: Comparison: Culture-directed Antibiotic vs Empiric Antibiotic; Test type: Superiority; p = .78, Chi-squared

6. Secondary Outcome: Monthly Enrollment Rate
Description: number of participants that were enrolled each month
Time Frame: Through study completion, an average of 17.5 months
Population: How many of the total 70 participants we enrolled per month
Measure: Median (Inter-Quartile Range); unit: participants enrolled per month
Groups:
- Monthly Enrollment Rate: Monthly Enrollment Rate (the number of patients on average enrolled per month to get to the total enrolled number)
Arm/Group | Monthly Enrollment Rate
Number analyzed (Participants) | 70
participants enrolled per month | 4 [2 to 5]

7. Secondary Outcome: Proportion of Enrolled Participants That Completed All Study Procedures
Description: Number of persons enrolled who completed all study procedures (completed all 4 follow-up questionnaires) divided by number participants enrolled
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Groups:
- Empiric Antibiotics: Antibiotic Protocol. For participants in the empiric Rx arm, we will choose an antibiotic with consideration of patient reported allergies, current medications and current Infectious Disease Society of American (IDSA) guidelines. If there is a contraindication to the first antibiotic on the list they will progress to the next option until a suitable selection is achieved.
  Antibiotics: Participants will be provided either nitrofurantoin 100 mg oral twice a day for 5 days, trimethoprim/sulfamethoxazole 875/125 oral twice a day for 3 days, fosfomycin 3g once oral, ciprofloxacin 250 mg oral twice a day for 5 days or cephalexin 500 mg oral twice a day for 5 days
Arm/Group | Culture-directed Antibiotic | Empiric Antibiotics
Number analyzed (Participants) | 35 | 35
Participants | 30 | 31
Statistical Analysis 1: Comparison: Culture-directed Antibiotic vs Empiric Antibiotics; Test type: Superiority; p = .78, Chi-squared

8. Secondary Outcome: Proportion of Enrolled Participants That Took Alternative Agents for Management of Symptoms
Description: Number of persons enrolled who took alternative agents for management of symptoms divided by number participants enrolled
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Culture-directed Antibiotic | Empiric Antibiotic
Number analyzed (Participants) | 35 | 35
Participants | 16 | 10
Statistical Analysis 1: Comparison: Culture-directed Antibiotic vs Empiric Antibiotic; Test type: Superiority; p = .68, Chi-squared

9. Secondary Outcome: Proportion of Participants in the Culture-directed Arm That Acquired Off-protocol Antibiotics for Their Symptoms
Description: Number of participants in the culture-directed arm that acquired off-protocol antibiotics for their symptoms divided by the number of participants in the culture-directed arm
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Groups:
- Culture-directed Arm: Culture-directed Arm of Participants Only
Arm/Group | Culture-directed Arm
Number analyzed (Participants) | 35
Participants | 1

10. Secondary Outcome: Proportion of Enrolled Participants That Completed Electronic Surveys
Description: Number of persons enrolled who completed all electronic surveys divided by number participants enrolled
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Culture-directed Antibiotic | Empiric Antibiotics
Number analyzed (Participants) | 35 | 35
Participants | 30 | 31
Statistical Analysis 1: Comparison: Culture-directed Antibiotic vs Empiric Antibiotics; Test type: Superiority; p = .78, Chi-squared

11. Other Pre Specified Outcome: Clinical Success at 14 Days
Description: Score of <1 on question 1 (urinary burning),3 (urinary urgency) and 5 (urinary frequency) on Urinary Tract Infection Symptom Assessment at day 14. A lower scale correlates with better symptoms with 0 being no symptoms and 1 being "little" symptoms.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Culture-directed Antibiotic | Empiric Antibiotic
Number analyzed (Participants) | 31 | 31
Participants | 19 | 12
Statistical Analysis 1: Comparison: Culture-directed Antibiotic vs Empiric Antibiotic; Test type: Superiority; p = 0.13, Chi-squared

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Culture-directed Antibiotic | Empiric Antibiotic
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 5/35 | 0/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Culture-directed Antibiotic (N=35) | Empiric Antibiotic (N=35)
Nausea/Vomiting Symptoms (Gastrointestinal disorders) | 3 (3) | 0 (0) — Nausea, vomiting
Diarrhea (Gastrointestinal disorders) | 5 (5) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT05726318/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/18/NCT05726318/ICF_001.pdf